CLINICAL TRIAL: NCT00560859
Title: A Randomized Controlled Study of Adenotonsillectomy for Children With Obstructive Sleep Apnea Syndrome
Brief Title: Childhood Adenotonsillectomy Study for Children With OSAS
Acronym: CHAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Harvard University (Other); University of Michigan (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 804695; 5U01HL083129-05 (NIH)
Record Dates: First submitted 2007-11-19; First posted 2007-11-20 (Estimated); Results first posted 2015-12-15 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-11

CONDITIONS: Obstructive Sleep Apnea; Snoring
Keywords: Sleep disordered breathing; Sleep apnea; Tonsillectomy; Adenoidectomy; Snoring; Neurobehavioral Manifestations; Obstructive Sleep Apnea Syndrome
MeSH Terms: conditions — Sleep Apnea, Obstructive; Snoring; Sleep Apnea Syndromes; Neurobehavioral Manifestations | interventions — Adenoidectomy; Watchful Waiting; Palliative Care

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early AT Surgery (Active Comparator): There will be removal of tonsils and adenoids that will be performed within 4 weeks of the baseline visit.
  Interventions: Procedure: Adenotonsillectomy (AT) - removal of adenoids and tonsils
- Watchful Waiting (Other): Children will be closely monitored and re-evaluated for AT by an otolaryngologist after the primary 7 month monitoring period.
  Interventions: Other: Watchful Waiting

INTERVENTIONS:
Procedure: Adenotonsillectomy (AT) - removal of adenoids and tonsils — Standard surgical intervention for treatment of Obstructive Sleep Apnea Syndrome which includes removal of adenoids and tonsils
  Other Names: EAT
  Arms: Early AT Surgery
Other: Watchful Waiting — Children will reevaluated for adenotonsillectomy (AT) after a 7 month primary monitoring period.
  Other Names: Watchful Waiting with Supportive Care (WWSC)
  Arms: Watchful Waiting

SUMMARY:
The purpose of this research is to determine the effect of adenotonsillectomy surgery (removal of tonsils and adenoids) on obstructive sleep apnea syndrome (OSAS) in children. OSAS can cause health problems including poor growth, high blood pressure, diabetes and behavioral and learning difficulties. Although adenotonsillectomy is the usual treatment for children with OSAS, it is not known with any certainty if the child's OSAS symptoms improve afterwards. This study will help determine if improvement occurs or if it does not. It will also look at whether certain groups, such as children who are overweight or of different ethnicities, are helped by the surgery.

DETAILED DESCRIPTION:
Because adenotonsillectomy is the usual treatment for OSAS, all children in the study will get surgery. However, in order to assess the extent to which adenotonsillectomy surgery improves breathing disturbances and sleep quality in children with OSAS, two groups will be studied. One group will get surgery early (one month after enrollment) and the other group will be re-evaluated for surgery within 7 months of enrollment.

Children in both groups will be closely monitored through the 7-8 month study period and sleep and health educational materials will be provided to assist in establishing healthy habits.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 5.0 to 9.99 years at time of screening.
2. Diagnosed with Obstructive Sleep Apnea defined as: Obstructive Apnea Index (OAI) ≥ 1 or Apnea Hypopnea Index (AHI) ≥ 2, confirmed on nocturnal, laboratory-based PSG and Parental report of habitual snoring (on average occurring >3 nights per week).
3. Tonsillar hypertrophy ≥ 1 based on a standardized scale of 0-4: 0 = surgically absent, 1 = taking up < 25% of the airway, 2 = 25 - 50 % of the airway,3 = 50 - 75 % of the airway, 4 = > 75% of the airway
4. Deemed to be a surgical candidate for AT by Ear, Nose and Throat specialist (ENT) evaluation.

Exclusion Criteria:

1. Recurrent tonsillitis defined as: >3 episodes in each of 3 years, 5 episodes in each of 2 years, or 7 episodes in one year
2. Craniofacial anomalies, including cleft lip and palate or sub-mucosal cleft palate or any anatomic or systemic condition which would interfere with general anesthesia or removal of tonsils and adenoid tissue in the standard fashion
3. Obstructive breathing while awake that merits prompt AT in the opinion of the child's physician
4. Severe OSAS or significant hypoxemia requiring immediate AT as defined by: OAI>20 or AHI>30, desaturation defined as oxygen saturation (SaO2) <90% for more than 2% sleep time
5. Apnea hypopnea indices in the normal range (OAI < 1 and AHI <2)
6. Evidence of clinically significant cardiac arrhythmia on PSG: Non-sustained ventricular tachycardia Atrial fibrillation, Second degree atrioventricular (AV) block: Sustained bradycardia < 40 bpm (> 2 minutes, Sustained tachycardia > 140 bpm (> 2 minutes)
7. Extremely overweight defined as: body mass index > 2.99 age group and sex-z-score
8. Severe health problems that could be exacerbated by delayed treatment for OSAS Including: Doctor-diagnosed heart disease or cor pulmonale, history of Stage II Hypertension (HTN) defined as > 99% percentile plus 5 mmHg for either systolic or diastolic, based on the age, gender, and height and/or requiring medication, therapy for failure to thrive or short stature, psychiatric or behavioral disorders requiring or likely to require initiation of new medication, therapy, or other specific treatment. School aged children, parental report of excessive daytime sleepiness defined as unable to maintain wakefulness, at least three times per week, in routine activities in school or home, despite adequate opportunity to sleep.
9. Severe chronic health conditions that might hamper participation including: severe cardiopulmonary disorders, sickle cell anemia, poorly controlled asthma, epilepsy requiring medication, diabetes (type I or type II) requiring medication, conditions likely to preclude accurate polysomnography (e.g. severe uncontrolled pain),mental retardation or enrollment in a formal school Individual Educational Plan (IEP) and assigned to a self-contained classroom for all academic subjects, history of inability to complete cognitive testing and/or score on the Differential Ability Scale (DAS) II of ≤ 55, chronic infection or HIV
10. Known genetic, craniofacial, neurological or psychiatric conditions likely to affect the airway, cognition, or behavior
11. Current use of one or more of the following medications: psychotropics, hypnotics,hypoglycemic agents or insulin,antihypertensives,growth hormone, anticonvulsants,anti-coagulants,daily oral corticosteroids, daily medications for pain
12. Previous upper airway surgery on the nose, pharynx or larynx, including tonsillectomy. Ear surgery and/or pressure equalizing (PE) tubes are not exclusion criteria
13. Receives Continuous Positive Airway Pressure (CPAP) treatment
14. A parent or guardian who cannot accompany the child on the night of polysomnogram (PSG)
15. A family planning to move out of the area within the year
16. Female participants only: Parental report that child has reached menarche

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 453 (Actual)
Dates: Start 2007-10; Primary Completion 2012-03 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Redline, MD, MPH, Study Chair — Harvard University; Susan Ellenberg, Ph.D., Study Director — University of Pennsylvania; Ron Chervin, MD, MS, Principal Investigator — University of Michigan; Bruno Giordani, PH.D., Study Director — Univeristy of Michigan; Susan Garetz, MD, Study Director — University of Michigan; Raouf Amin, MD, Principal Investigator — Cincinnati Children's Hopsital Medical Center (CCHMC); Carole Marcus, MBB Ch., Principal Investigator — Children's Hospital of Philadelphia; Carol Rosen, MD, Principal Investigator — Case University School of Medicine; Rainbow Babies & Children's Hospital; Ron Mitchell, MD, Principal Investigator — Cardinal Glennon Children's Medical Center, St. Louis MO; Raanan Arens, MD, Principal Investigator — Montefiore Children's Hospital Albert Einstein Med Ctr, NY NY; Hiren Muzumdar, MD, Principal Investigator — Montefiore Chilren's Hospital Albert Einstein Med Ctr, NY NY; Eliot Katz, MD, Principal Investigator — Boston Children's Hospital, Boston MA
Locations (6):
- United States (6):
  - Children's Hospital Boston, Boston, Massachusetts
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Montefiore Children's Hospital, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies & Children's Hospital, Cleveland, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Tsou PY, Alex RM, Redline S, Sands SA. Pathophysiological Traits in Pediatric Obstructive Sleep Apnea. Associations with Patient Characteristics and Responses to Therapy: A Secondary Analysis of the CHAT Clinical Trial. Ann Am Thorac Soc. 2025 Dec;22(12):1931-1941. doi: 10.1513/AnnalsATS.202412-1302OC. PMID 40720163
- [Derived] Ramirez-Contreras C, Elgueta VP, Briones-Suarez L. Childhood OSAS and Obesity: Prospective Associations of Anthropometric Markers With Objective Sleep Outcomes in the CHAT Trial. J Sleep Res. 2025 Jul 17:e70156. doi: 10.1111/jsr.70156. Online ahead of print. PMID 40676770
- [Derived] Dai S, Yang M, Au CT, Yuen NTK, Zhang Y, Tang A, Yu MWL, Li AM, Chan KCC. Supine position-related obstructive sleep apnea in children: insights from the Childhood Adenotonsillectomy Trial. Sleep Breath. 2025 Jun 30;29(4):230. doi: 10.1007/s11325-025-03393-1. PMID 40587023
- [Derived] Wang C, Sun K, Liu K, Yu Z. Association of allergic rhinitis with persistent obstructive sleep apnea: A secondary analysis of the childhood adenotonsillectomy trial. Sleep Med. 2024 Mar;115:246-250. doi: 10.1016/j.sleep.2024.02.029. Epub 2024 Feb 15. PMID 38382311
- [Derived] Wang C, Hu H, Sun K, Ma Y, Lu Y, Liu K, Yu Z. Dysphagia Outcomes Before and After Adenotonsillectomy in Children With Obstructive Sleep Apnea: A Secondary Analysis of a Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2023 Oct 1;149(10):878-883. doi: 10.1001/jamaoto.2023.2145. PMID 37590002
- [Derived] Williamson AA, Fan J, Distel L, Xiao R, Stefanovski D, Tapia IE. Nighttime sleep duration and variability in children with obstructive sleep apnea syndrome: Sociodemographic disparities and neurobehavioral outcomes. Sleep Med. 2023 Feb;102:165-172. doi: 10.1016/j.sleep.2023.01.003. Epub 2023 Jan 10. PMID 36682144
- [Derived] Magnusdottir S, Witmans M, Hilmisson H. Sleep quality, sleep apnea, and metabolic health in children treated with adenotonsillectomy. Sleep Breath. 2023 Aug;27(4):1527-1540. doi: 10.1007/s11325-022-02747-3. Epub 2022 Nov 24. PMID 36434376
- [Derived] Yu PK, Radcliffe J, Gerry Taylor H, Amin RS, Baldassari CM, Boswick T, Chervin RD, Elden LM, Furth SL, Garetz SL, George A, Ishman SL, Kirkham EM, Liu C, Mitchell RB, Kamal Naqvi S, Rosen CL, Ross KR, Shah JR, Tapia IE, Young LR, Zopf DA, Wang R, Redline S. Neurobehavioral morbidity of pediatric mild sleep-disordered breathing and obstructive sleep apnea. Sleep. 2022 May 12;45(5):zsac035. doi: 10.1093/sleep/zsac035. Epub 2022 Feb 12. PMID 35554583
- [Derived] Snow A, Vazifedan T, Baldassari CM. Evaluation of Nocturnal Enuresis After Adenotonsillectomy in Children With Obstructive Sleep Apnea: A Secondary Analysis of a Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2021 Oct 1;147(10):887-892. doi: 10.1001/jamaoto.2021.2303. PMID 34499109
- [Derived] Martin-Montero A, Gutierrez-Tobal GC, Kheirandish-Gozal L, Vaquerizo-Villar F, Alvarez D, Del Campo F, Gozal D, Hornero R. Heart rate variability as a potential biomarker of pediatric obstructive sleep apnea resolution. Sleep. 2022 Feb 14;45(2):zsab214. doi: 10.1093/sleep/zsab214. PMID 34498074
- [Derived] Isaiah A, Spanier AJ, Grattan LM, Wang Y, Pereira KD. Predictors of Behavioral Changes After Adenotonsillectomy in Pediatric Obstructive Sleep Apnea: A Secondary Analysis of a Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2020 Oct 1;146(10):900-908. doi: 10.1001/jamaoto.2020.2432. PMID 32880655
- [Derived] Hartmann S, Bruni O, Ferri R, Redline S, Baumert M. Cyclic alternating pattern in children with obstructive sleep apnea and its relationship with adenotonsillectomy, behavior, cognition, and quality of life. Sleep. 2021 Jan 21;44(1):zsaa145. doi: 10.1093/sleep/zsaa145. PMID 32777055
- [Derived] Hilmisson H, Berman S, Magnusdottir S. Sleep apnea diagnosis in children using software-generated apnea-hypopnea index (AHI) derived from data recorded with a single photoplethysmogram sensor (PPG) : Results from the Childhood Adenotonsillectomy Study (CHAT) based on cardiopulmonary coupling analysis. Sleep Breath. 2020 Dec;24(4):1739-1749. doi: 10.1007/s11325-020-02049-6. Epub 2020 Mar 28. PMID 32222900
- [Derived] Isaiah A, Pereira KD, Das G. Polysomnography and Treatment-Related Outcomes of Childhood Sleep Apnea. Pediatrics. 2019 Oct;144(4):e20191097. doi: 10.1542/peds.2019-1097. PMID 31533972
- [Derived] Hilmisson H, Lange N, Magnusdottir S. Objective sleep quality and metabolic risk in healthy weight children results from the randomized Childhood Adenotonsillectomy Trial (CHAT). Sleep Breath. 2019 Dec;23(4):1197-1208. doi: 10.1007/s11325-019-01802-w. Epub 2019 Feb 23. PMID 30798410
- [Derived] Hodges E, Marcus CL, Kim JY, Xanthopoulos M, Shults J, Giordani B, Beebe DW, Rosen CL, Chervin RD, Mitchell RB, Katz ES, Gozal D, Redline S, Elden L, Arens R, Moore R, Taylor HG, Radcliffe J, Thomas NH. Depressive symptomatology in school-aged children with obstructive sleep apnea syndrome: incidence, demographic factors, and changes following a randomized controlled trial of adenotonsillectomy. Sleep. 2018 Dec 1;41(12):zsy180. doi: 10.1093/sleep/zsy180. PMID 30212861
- [Derived] Liu X, Immanuel S, Kennedy D, Martin J, Pamula Y, Baumert M. Effect of adenotonsillectomy for childhood obstructive sleep apnea on nocturnal heart rate patterns. Sleep. 2018 Nov 1;41(11):zsy171. doi: 10.1093/sleep/zsy171. PMID 30165465
- [Derived] Thomas NH, Xanthopoulos MS, Kim JY, Shults J, Escobar E, Giordani B, Hodges E, Chervin RD, Paruthi S, Rosen CL, Taylor GH, Arens R, Katz ES, Beebe DW, Redline S, Radcliffe J, Marcus CL. Effects of Adenotonsillectomy on Parent-Reported Behavior in Children With Obstructive Sleep Apnea. Sleep. 2017 Apr 1;40(4):zsx018. doi: 10.1093/sleep/zsx018. PMID 28199697
- [Derived] Liu X, Immanuel S, Pamula Y, Kennedy D, Martin J, Baumert M. Adenotonsillectomy for childhood obstructive sleep apnoea reduces thoraco-abdominal asynchrony but spontaneous apnoea-hypopnoea index normalisation does not. Eur Respir J. 2017 Jan 25;49(1):1601177. doi: 10.1183/13993003.01177-2016. Print 2017 Jan. PMID 27811072
- [Derived] Wang R, Dong Y, Weng J, Kontos EZ, Chervin RD, Rosen CL, Marcus CL, Redline S. Associations among Neighborhood, Race, and Sleep Apnea Severity in Children. A Six-City Analysis. Ann Am Thorac Soc. 2017 Jan;14(1):76-84. doi: 10.1513/AnnalsATS.201609-662OC. PMID 27768852
- [Derived] Paruthi S, Buchanan P, Weng J, Chervin RD, Mitchell RB, Dore-Stites D, Sadhwani A, Katz ES, Bent J, Rosen CL, Redline S, Marcus CL. Effect of Adenotonsillectomy on Parent-Reported Sleepiness in Children with Obstructive Sleep Apnea. Sleep. 2016 Nov 1;39(11):2005-2012. doi: 10.5665/sleep.6232. PMID 27568804
- [Derived] Taylor HG, Bowen SR, Beebe DW, Hodges E, Amin R, Arens R, Chervin RD, Garetz SL, Katz ES, Moore RH, Morales KH, Muzumdar H, Paruthi S, Rosen CL, Sadhwani A, Thomas NH, Ware J, Marcus CL, Ellenberg SS, Redline S, Giordani B. Cognitive Effects of Adenotonsillectomy for Obstructive Sleep Apnea. Pediatrics. 2016 Aug;138(2):e20154458. doi: 10.1542/peds.2015-4458. PMID 27464674
- [Derived] Paruthi S, Rosen CL, Wang R, Weng J, Marcus CL, Chervin RD, Stanley JJ, Katz ES, Amin R, Redline S. End-Tidal Carbon Dioxide Measurement during Pediatric Polysomnography: Signal Quality, Association with Apnea Severity, and Prediction of Neurobehavioral Outcomes. Sleep. 2015 Nov 1;38(11):1719-26. doi: 10.5665/sleep.5150. PMID 26414902
- [Derived] Chervin RD, Ellenberg SS, Hou X, Marcus CL, Garetz SL, Katz ES, Hodges EK, Mitchell RB, Jones DT, Arens R, Amin R, Redline S, Rosen CL; Childhood Adenotonsillectomy Trial. Prognosis for Spontaneous Resolution of OSA in Children. Chest. 2015 Nov;148(5):1204-1213. doi: 10.1378/chest.14-2873. PMID 25811889
- [Derived] Quante M, Wang R, Weng J, Rosen CL, Amin R, Garetz SL, Katz E, Paruthi S, Arens R, Muzumdar H, Marcus CL, Ellenberg S, Redline S; Childhood Adenotonsillectomy Trial (CHAT). The Effect of Adenotonsillectomy for Childhood Sleep Apnea on Cardiometabolic Measures. Sleep. 2015 Sep 1;38(9):1395-403. doi: 10.5665/sleep.4976. PMID 25669177
- [Derived] Garetz SL, Mitchell RB, Parker PD, Moore RH, Rosen CL, Giordani B, Muzumdar H, Paruthi S, Elden L, Willging P, Beebe DW, Marcus CL, Chervin RD, Redline S. Quality of life and obstructive sleep apnea symptoms after pediatric adenotonsillectomy. Pediatrics. 2015 Feb;135(2):e477-86. doi: 10.1542/peds.2014-0620. Epub 2015 Jan 19. PMID 25601979
- [Derived] Mitchell RB, Garetz S, Moore RH, Rosen CL, Marcus CL, Katz ES, Arens R, Chervin RD, Paruthi S, Amin R, Elden L, Ellenberg SS, Redline S. The use of clinical parameters to predict obstructive sleep apnea syndrome severity in children: the Childhood Adenotonsillectomy (CHAT) study randomized clinical trial. JAMA Otolaryngol Head Neck Surg. 2015 Feb;141(2):130-6. doi: 10.1001/jamaoto.2014.3049. PMID 25474490
- [Derived] Katz ES, Moore RH, Rosen CL, Mitchell RB, Amin R, Arens R, Muzumdar H, Chervin RD, Marcus CL, Paruthi S, Willging P, Redline S. Growth after adenotonsillectomy for obstructive sleep apnea: an RCT. Pediatrics. 2014 Aug;134(2):282-9. doi: 10.1542/peds.2014-0591. PMID 25070302
- [Derived] Weinstock TG, Rosen CL, Marcus CL, Garetz S, Mitchell RB, Amin R, Paruthi S, Katz E, Arens R, Weng J, Ross K, Chervin RD, Ellenberg S, Wang R, Redline S. Predictors of obstructive sleep apnea severity in adenotonsillectomy candidates. Sleep. 2014 Feb 1;37(2):261-9. doi: 10.5665/sleep.3394. PMID 24497655
- [Derived] Marcus CL, Moore RH, Rosen CL, Giordani B, Garetz SL, Taylor HG, Mitchell RB, Amin R, Katz ES, Arens R, Paruthi S, Muzumdar H, Gozal D, Thomas NH, Ware J, Beebe D, Snyder K, Elden L, Sprecher RC, Willging P, Jones D, Bent JP, Hoban T, Chervin RD, Ellenberg SS, Redline S; Childhood Adenotonsillectomy Trial (CHAT). A randomized trial of adenotonsillectomy for childhood sleep apnea. N Engl J Med. 2013 Jun 20;368(25):2366-76. doi: 10.1056/NEJMoa1215881. Epub 2013 May 21. PMID 23692173
- See also: National Center on Sleep Disorder Research — http://www.nhlbi.nih.gov/about/ncsdr/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Children were recruited at 7 academic sleep centers. Early in the trial the investigator at one center relocated and that center was withdrawn.
Groups:
- Early AT Surgery: Adenotonsillectomy (AT) - removal of tonsils and adenoids - performed within 4 weeks of the baseline visit.
  Adenotonsillectomy (AT) - removal of adenoids and tonsils: Standard surgical intervention for treatment of Obstructive Sleep Apnea Syndrome.
- Watchful Waiting: Children will be closely monitored during the primary 7 month monitoring period and will be re-evaluated for AT by an otolaryngologist at the end of that period. a
  Watchful Waiting: Children will reevaluated for adenotonsillectomy (AT) after a 7 month primary monitoring period.
Period: Overall Study
Arm/Group | Early AT Surgery | Watchful Waiting
Started | 226 | 227
Completed | 194 | 203
Not Completed | 32 | 24

BASELINE CHARACTERISTICS:
Population: These numbers represent all children randomized .
Groups:
- Total: Total of all reporting groups
Arm/Group | Early AT Surgery | Watchful Waiting | Total
Number analyzed (Participants) | 226 | 227 | 453
Age, Continuous [Mean (Standard Deviation); unit: Years] | 6.6 (1.4) | 6.5 (1.4) | 6.6 (1.4)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 226 | 227 | 453
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 125 | 109 | 234
  Male | 101 | 118 | 219
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 126 | 123 | 249
  White | 74 | 81 | 155
  More than one race | 15 | 12 | 27
  Unknown or Not Reported | 6 | 6 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 21 | 37
  Not Hispanic or Latino | 210 | 206 | 416
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 226 | 227 | 453

OUTCOME MEASURES:

1. Primary Outcome: Improvements in Attention/Executive Domain Index of the Developmental Neuropsychological Assessment (NEPSY) From Baseline to 7 Months.
Description: The primary outcome was the change in the attention and executive function score on the NEPSY. The change from baseline in Attention/Executive Domain Index of the Developmental Neuropsychological Assessment (NEPSY) was compared to 7 months were compared. Scores on the attention and executive-function domain of the Developmental Neuropsychological Assessment (NEPSY) range from 50 to 150, with higher scores indicating better functioning.
Time Frame: The primary endpoint measure will occur at 7 months following the baseline visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Watchful Waiting: Children will be closely monitored during the primary 7-month monitoring period and re-evaluated for AT by an otolaryngologist after that period.
  Watchful Waiting: Children will reevaluated for adenotonsillectomy (AT) after a 7 month primary monitoring period.
Arm/Group | Early AT Surgery | Watchful Waiting
Number analyzed (Participants) | 194 | 203
units on a scale | 7.1 (13.9) | 5.1 (13.4)
Statistical Analysis 1: Comparison: Early AT Surgery vs Watchful Waiting; Test type: Superiority or Other; p = 0.16, ANCOVA; difference of change from baseline = 2.0

2. Secondary Outcome: Change in Apnea Hypopnea Index (AHI) Score From Baseline to 7 Months
Description: The outcome measure was the change in AHI from baseline to 7 months to determine if there was an improvement in score is associated with improved OSAS (i.e reduction in AHI). The AHI is calculated by dividing the number of apnea events by the number of hours of sleep. The obstructive sleep apnea syndrome was defined as an AHI score of 2 or more events per hour or an obstructive apnea index (OAI) score of 1 or more events per hour.
Time Frame: 7 months following the baseline visit.
Measure: Median (Inter-Quartile Range); unit: Events per hour
Arm/Group | Early AT Surgery | Watchful Waiting
Number analyzed (Participants) | 194 | 203
Events per hour | -3.5 [-7.1 to -1.8] | -1.6 [-3.7 to 0.5]

3. Secondary Outcome: Change in Score of Pediatric Sleep Questionnaire Sleep-related Breathing Disorder Scale
Description: Scores on the Pediatric Sleep Questionnaire sleep-related breathing disorder scale (PSQ-SRBD) range from 0 to 1, with higher scores indicating greater severity.
Time Frame: 7 months following baseline.
Population: There was missing data for some children in the Watchful Waiting group since the Pediatric Sleep Questionnaire was not completed. Hence these numbers are not consistent with the rows in the participant flow module
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Early AT Surgery | Watchful Waiting
Number analyzed (Participants) | 194 | 202
units on a scale | -0.3 (0.2) | 0 (0.2)

ADVERSE EVENTS:
Time Frame: Reported adverse events include events starting from the initiation of any study procedures to the end of the study follow-up.
Arm/Group | Early AT Surgery | Watchful Waiting
Serious Adverse Events (participants affected / at risk) | 7/226 | 9/227
Other Adverse Events (participants affected / at risk) | 166/226 | 227/227
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Early AT Surgery (N=226) | Watchful Waiting (N=227)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Application site pain (General disorders) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Pleural Effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tonsillar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Hypersomnia (Nervous system disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Vomitting (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Early AT Surgery (N=226) | Watchful Waiting (N=227)
Abdominal Discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute Sinusitis (Infections and infestations) | 3 (3) | 2 (2)
Adenoviral upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
Allergic cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Allergy to sting (Immune system disorders) | 0 (0) | 1 (1)
Animal Bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ankle Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Application site bleeding (General disorders) | 1 (1) | 0 (0)
Application site rash (General disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 14 (14)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Attention Deficit/Hyperactivitiy disorder (Psychiatric disorders) | 3 (3) | 4 (4)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Blood Glucose (Investigations) | 0 (0) | 1 (1)
Body Tinea (Infections and infestations) | 1 (1) | 1 (1)
Breath Odor (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 3 (3)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Choking sensation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Conjuctivits (Eye disorders) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 15 (15) | 11 (11)
Croup Infectious (Infections and infestations) | 0 (0) | 1 (1)
Croup Non infectious (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diabetes Mellitus non-insulin dependent (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ear Infection (Infections and infestations) | 4 (4) | 8 (8)
Ear Infection Baceterial (Infections and infestations) | 7 (7) | 4 (4)
Ear Pain (Ear and labyrinth disorders) | 3 (3) | 2 (2)
Ear Piercing (Social circumstances) | 1 (1) | 0 (0)
Ear Tube removal (Surgical and medical procedures) | 0 (0) | 1 (1)
electroencephalogram abnormal (Investigations) | 1 (1) | 1 (1)
Emergency care examination normal (Investigations) | 1 (1) | 0 (0)
Enuresis (Renal and urinary disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
External ear infection (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Eye Allergy (Eye disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
fatigue (General disorders) | 0 (0) | 1 (1)
Febrile infection (Infections and infestations) | 2 (2) | 1 (1)
fever (in the absence of neutropenia, where neutropenia is defined as anc <1.0 x 10e9/l) (General disorders) | 0 (0) | 1 (1)
Finger nail removal (Surgical and medical procedures) | 0 (0) | 1 (1)
Foreign body in eye (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis adenovirus (Infections and infestations) | 0 (0) | 1 (1)
gastroenteritis viral (Infections and infestations) | 1 (1) | 4 (4)
gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0)
genital rash (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Growing pains (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Hand-foot-and-mouth disease (Infections and infestations) | 1 (1) | 1 (1)
head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
headache (Nervous system disorders) | 1 (1) | 6 (6)
Heart rate irregular (Investigations) | 0 (0) | 1 (1)
hordeolum (Infections and infestations) | 0 (0) | 1 (1)
hypersomnia (Nervous system disorders) | 1 (1) | 0 (0)
incision site pain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
infected insect bite (Infections and infestations) | 2 (2) | 1 (1)
infection with unknown anc - bladder (urinary) (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
influenza (Infections and infestations) | 2 (2) | 3 (3)
influenza like illness (General disorders) | 0 (0) | 4 (4)
laceration (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Lice infestation (Infections and infestations) | 0 (0) | 1 (1)
loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
multiple allergies (Immune system disorders) | 0 (0) | 1 (1)
muscle injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Nail Tinea (Infections and infestations) | 1 (1) | 0 (0)
nasal cavity/paranasal sinus reactions (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 10 (10)
nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 6 (6) | 4 (4)
Otitis media bacterial (Infections and infestations) | 0 (0) | 1 (1)
pain management (Surgical and medical procedures) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 4 (4) | 7 (7)
pharyngitis streptococcal (Infections and infestations) | 2 (2) | 5 (5)
pneumonia (Infections and infestations) | 4 (4) | 2 (2)
pneumonia mycoplasmal (Infections and infestations) | 1 (1) | 1 (1)
post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
postoperative fever (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
precocious puberty (Endocrine disorders) | 1 (1) | 0 (0)
productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
pyrexia (General disorders) | 1 (1) | 0 (0)
rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
relapsing fever (Infections and infestations) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 2 (2)
Rhinitis seasonal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinovirus infection (Infections and infestations) | 0 (0) | 1 (1)
road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Scarlet Fever (Infections and infestations) | 0 (0) | 2 (2)
Seasonal Allergy (Immune system disorders) | 2 (2) | 4 (4)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Sinus headache (Nervous system disorders) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Sleep Apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5)
Snoring (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Staphylococcal skin infection (Infections and infestations) | 1 (1) | 0 (0)
Stomach discomfort (Gastrointestinal disorders) | 0 (0) | 2 (2)
Streptococcal bacteraemia (Infections and infestations) | 4 (4) | 6 (6)
Streptococcal infection (Infections and infestations) | 3 (3) | 8 (8)
Sweating fever (Infections and infestations) | 2 (2) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
Tinea infection (Infections and infestations) | 1 (1) | 0 (0)
Tongue Tie operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Tonsillar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 2 (2)
Tonsillitis streptococcal (Infections and infestations) | 0 (0) | 2 (2)
Tooth Infection (Infections and infestations) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Torticollis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tympanometry (Investigations) | 0 (0) | 1 (1)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 10 (10)
Upper respiratory tract infection (Infections and infestations) | 6 (6) | 3 (3)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 4 (4)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Varicella (Infections and infestations) | 0 (0) | 1 (1)
vasomotor rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Viral Infection (Infections and infestations) | 1 (1) | 2 (2)
Viral Rash (Infections and infestations) | 1 (1) | 0 (0)
Viral Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Viral Upper Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Vomitting (Gastrointestinal disorders) | 3 (3) | 4 (4)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Children under 5 years of age, in whom OSAS is common, were not included. Children on medications for ADHD or with prolonged oxygen-hemoglobin desaturation were also excluded, so results cannot be extrapolated to such children.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No